CLINICAL TRIAL: NCT07152795
Title: Weizmannia Coagulans BC99 Improved Intestinal Motility and Chronic Constipation Through Regulating Gut Microbiota: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Probiotics for Alleviating Chronic Constipation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20250825
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): Participants receive one sachet per day containing probiotic BC99 and maltodextrin (Week 0 to Week8).
  Interventions: Dietary Supplement: Probiotic
- Placebo Group (Placebo Comparator): Participants receive one sachet per day containing maltodextrin only, serving as the placebo(Week 0 to Week8).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — During the intervention, participants can consume BC99 daily and any adverse reactions were noted. Stool and serum samples were collected for analysis of 16S rRNA and serum inflammatory markers. Changes in intestinal flora and inflammatory factors before and after supplementation were assessed.
  Arms: Probiotic Group
Dietary Supplement: Placebo — During the intervention, participants can consume maltodextrin daily and any adverse reactions were noted. Stool and serum samples were collected for analysis of 16S rRNA and serum inflammatory markers. Changes in intestinal flora and inflammatory factors before and after supplementation were assessed.
  Arms: Placebo Group

SUMMARY:
To investigate the clinical effects of probiotics in relieving intestinal motility and chronic constipation through regulating gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults aged 18-70 years who meet the Rome IV diagnostic criteria for chronic constipation (duration of at least 6 months, with less than 3 bowel movements per week and/or Bristol Stool Scale types 1 and 2);
2. Not using laxatives rarely leads to loose stools；
3. The standard for irritable bowel syndrome is insufficient;
4. Research participants (including male subjects) who have no family planning within 14 days prior to screening and voluntarily take effective contraceptive measures within 6 months after the end of the trial;
5. Patients capable of understanding the clinical study and willing to comply with the study requirements and procedures;
6. Subjects who have signed the informed consent form. -

Exclusion Criteria:

(1) The use of probiotics, prebiotics, or antibiotics within 2 weeks of enrollment; (2) Regular use of a high-fiber diet, as measured by the recommended food score (RFS); (3) Regular use of medications affecting bowel habits, such as irritable bowel syndrome, functional bloating, and functional diarrhea; (4) Currently have, or have had in the past 2 years, any gastrointestinal conditions such as: Crohn's disease, celiac disease, Ulcerative colitis, Malignant tumor of the colon; (5) Medical history of cardiovascular, liver, or renal diseases; alcoholics; (6) Hypersensitivity to probiotics or the ingredients used in this study; (7) Pregnancy or breastfeeding; (8) Participation in another clinical trial in the 3 months before enrollment.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Assessing the Improvement of Chronic Constipation Symptoms Following Probiotic Intervention. | 8 weeks
  Constipation symptoms are measured using Bristol Stool Form Scale, where 1 and 2 indicate constipation with hard stools, 3 and 4 show normal conditions with ideal stool form, and 5, 6, and 7 suggest diarrhea with stools becoming softer to watery.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan University of Science and Technolog, Luoyang, Henan, China